CLINICAL TRIAL: NCT02151396
Title: Effect of Working Memory Training on ADHD Brain Function
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hartford Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: R21HD061915 (NIH)
Record Dates: First submitted 2014-05-28; First posted 2014-05-30 (Estimated); Last update posted 2014-05-30 (Estimated); Status verified 2014-05

CONDITIONS: Attention-Deficit/Hyperactivity Disorder (Combined-subtype)
Keywords: ADHD, hyperactivity, inattention, working memory
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Spasm | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cogmed Working Memory Training (Experimental): Cogmed (TM) working memory training following standard, recommended administration procedures
  Interventions: Behavioral: Working memory training; Device: Functional magnetic resonance imaging (fMRI)

INTERVENTIONS:
Behavioral: Working memory training
Device: Functional magnetic resonance imaging (fMRI)

SUMMARY:
There is evidence both that computer-administered cognitive training can improve ADHD working memory deficits and that this type of training in non-ADHD enhances normal working memory ability by altering brain activity in prefrontal cortex and the parietal lobe. However, no study has characterized brain activity changes following working memory training in ADHD to understand what neural changes occur when cognitive deficits are remedied. This R21 exploratory study will examine the neural basis of cognitive training treatment gains in working memory, ADHD symptoms, and various other executive abilities. We will test the hypothesis that working memory training increases frontoparietal brain activation and examine other regions to see if there is any evidence for "neural compensation" (i.e., engagement of brain regions after training that are not normally recruited for task performance).

DETAILED DESCRIPTION:
There is evidence both that computer-administered cognitive training can improve ADHD working memory deficits and that this type of training in non-ADHD enhances normal working memory ability by altering brain activity in prefrontal cortex and the parietal lobe. However, no study has characterized brain activity changes following working memory training in ADHD to understand what neural changes occur when cognitive deficits are remedied. This R21 exploratory study will examine the neural basis of cognitive training treatment gains in working memory, ADHD symptoms, and various other executive abilities. The study will compare n=21 ADHD adolescents with evidence for baseline deficits in working memory (i.e., <1.5 SD below normative ratings at baseline) before and after working memory training. Participants will undergo baseline neuropsychological and fMRI imaging with verbal and visuospatial Sternberg fMRI working memory tasks, 5 weeks of daily computerized working memory training, and then endpoint fMRI and cognitive evaluation of neural and behavioral changes. Training will utilize commercially-available Cogmed software (http://www.cogmed.com) as it has a well-developed set of computerized tools, with numerous practical advantages for this study. Our analyses will identify which brain regions in ADHD adolescents are affected by working memory treatment and characterize patterns of activation change between baseline and endpoint. We will examine post-treatment differences in the extent of activation and functional connectivity among activated brain regions to test hypotheses about possible neural mechanisms underlying treatment gains. Finally, we will conduct a series of analyses to determine what changes in brain function underlie a generalized effect of working memory training on ADHD symptoms and other 'executive' abilities. By identifying the neural correlates any such effect, this study could yield invaluable information about what the neural targets of any effective ADHD treatment must be. The key accomplishment of this exploratory study will be to characterize the neural basis of treatment gains in ADHD by testing theoretically-guided hypotheses about possible neuroplastic changes. The results will support larger, future studies aimed at better understanding the neural basis of this alternative treatment for ADHD, identifying biological or genetic factors that might denote the presence of a remediable working memory deficit, and ultimately achieving a better understanding of the etiology of ADHD working memory deficits.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be 13-17 years old and >6th grade English reading level to complete self-report evaluations (most are only available in English). ADHD-C participants must meet DSM-IV criteria (314.01).

Exclusion Criteria:

* Head injury sufficient to have caused >30 minutes lost consciousness; past or current CNS disease (e.g. stroke, MS, epilepsy or any repeated seizure history, tumor, etc) or brain lesion identified by MR (structural MR scans will be reviewed by a radiologist for the presence of clinical neuropathology that may affect cognitive task performance); Axis I DSM-IV lifetime history Bipolar disorder, psychotic disorder, OCD, PTSD, Tourette's disorder, Pervasive developmental disorder (e.g., Autistic disorder, PDD NOS, etc.); current DSM-IV substance dependence, Major Depressive Disorder or anxiety disorder; hypertension or juvenile-onset diabetes (current treatment with antihypertensives or insulin); current pregnancy (menstruating females will be tested); IQ estimate <80; left-handedness; psychotropic medication other than common psychostimulants that act primarily on dopamine neurotransmission systems. For instance, ADHD-C medications such as Wellbutrin (Buproprion), Strattera (Atomoxetine HCl), Cylert (Pemoline), or Provigil (Modafinil) will exclude participation; report of psychotic illness in first degree relative. Note, current DSM-IV disorders serve as exclusionary criteria to avoid the possibility of acute brain activity differences related more greatly to these disorders than ADHD. These stringent exclusion criteria are an advantage over many previous ADHD studies. However, given the frequent comorbidity and suspected biological liability among ADHD, substance, mood, and anxiety disorders, a lifetime history of mood or anxiety disorders will not exclude participation. Likewise, the frequent occurrence of CD/ODD and specific learning disabilities will not exclude participation.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 37 (Actual)
Dates: Start 2009-07; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Functional magnetic resonance imaging (fMRI) | 5 weeks
  fMRI assessment of working memory-related brain function

SECONDARY OUTCOMES:
Working memory neuropsychological test performance | 5 weeks
  Several tests of working memory abillity
ADHD clinical dysfunction | 5 weeks
  Parent- and self-reported ADHD symptom severity, ADHD-related problems, and role impairment at home

CONTACTS AND LOCATIONS:
Overall Officials: Michael C. Stevens, Ph.D., Principal Investigator — Hartford Hospital
Locations (1):
- Olin Neurospychiatry Research Center, Hartford, Connecticut, United States